CLINICAL TRIAL: NCT02874196
Title: Study of Diagnostic Performances of Dual Energy Imaging With Flat Detectors and Tomosynthesis in Identification of Loosening of Painful Hip Prosthesis
Brief Title: Prosthesis Loosening Imaging With Dual Energy and Tomosynthesis
Acronym: PLIDET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00677-34
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Hip Prosthesis Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with painful prosthesis (Experimental)
  Interventions: Procedure: Standard arthrography; Procedure: Dual energy arthrography; Procedure: Arthro-tomosynthesis; Procedure: Arthro-tomography; Procedure: Surgery on painful prosthesis

INTERVENTIONS:
Procedure: Standard arthrography
Procedure: Dual energy arthrography
Procedure: Arthro-tomosynthesis
Procedure: Arthro-tomography
Procedure: Surgery on painful prosthesis — Possibly performed during 6 months from arthrography

SUMMARY:
The purpose is to determine diagnostic performances of flat panel dual energy arthrography and arthro-tomosynthesis in identification of loosening of painful hip prosthesis, taking as reference the results of surgery performed 6 months after arthrography.

Secondary purposes are:

* To describe the level of concordance of each technique with the indication for surgery
* To study inter-technique concordance with kappa coefficient
* To study the relationship between density differential between 2 acquisitions and grey level on subtraction, i.e. subtraction quality according to metal

DETAILED DESCRIPTION:
Hip arthroplasty has become one of the most performed orthopedic procedures. Actual average lifetime of total hip prosthesis is approximately 15 years. Some complications are inevitable. Total hip prosthesis imaging, performed to search for a complication or wear, is difficult and depends on many techniques. Subtracted arthrography is a good technique but its access is limited because it needs an angiography room.

In this study patients undergo standard arthrography, dual energy arthrography, arthro-tomosynthesis and arthro-tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients sent for arthro-tomography of painful prosthesis, without contraindications to arthrography or injection of contrast agent
* Aware and cooperative
* Signed informed consent
* Affiliation to social security

Exclusion Criteria:

* Any contraindication to arthrography or injection of contrast agent
* Pregnant or possibly pregnant women
* Patient under guardianship
* Refusal or impossibility of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence or absence of prosthesis loosening detected with 3 radiographic techniques (dual-energy arthrography, arthro-tomosynthesis and single-energy tomography) and surgery | from day 0 up to 6 months
  Gold standard is presence or absence of prosthesis loosening revealed with surgery performed after 6 months from arthrography.
  Data of patients undergone surgery and not are collected and analyzed. Any clinical or imagery sign of loosening in non-operated patient, will be classified as loosening. A surgery decision for suspicion of loosening will be considered loosening.

SECONDARY OUTCOMES:
Comparison between density differential between 2 acquisitions and grey level on subtraction | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Alain Blum, Principal Investigator — Service d'Imagerie Guilloz - CHU Nancy - France
Locations (2):
- France (2):
  - CHU de Nancy, Nancy
  - SINCAL, Nancy

IPD SHARING:
Plan to Share IPD: No